CLINICAL TRIAL: NCT00220610
Title: Right Parietal Inhibition With rTMS in the Treatment of Depression
Brief Title: REPETITIVE TRANSCRANIAL MAGNETIC STIMULATION IN the Treatment of DEPRESSION
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Lucas Andreas Ziekenhuis Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCMO03.3741/SH/P03.1231L
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2005-09-22 (Estimated); Status verified 2005-09

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial magnetic stimulation

SUMMARY:
Subjects received rTMS daily on 10 consecutive weekdays (five sessions per week), during 20 minutes per session.During the rTMS session, the coil was centered flat over the right parietal cortex.

We follow the patient during 12 weeks after the 2 weeks of tms (follow-up period) to measure the depression with different rating scales.

We hypothesized that rTMS has a positive effect in the treatment of depression

ELIGIBILITY:
Inclusion Criteria:

* In and outpatients aged between 16 and 65 who met DSM-IV criteria for major depressive episode, and who had a score of 25 or higher on the 10-item Montgomery Asberg Depression Rating Scale (MADRS) were included

Exclusion Criteria:

* A history of epilepsy and any other medical disorder that should preclude the administration of rTMS. Only SSRI's, Mirtazapine and Promethazine as psychotropic medication was accepted if the dosage of antidepressive medication had not been changed for 6 weeks, and if the dosage of Promethazine had not been changed for 2 weeks prior to inclusion. Antidepressive medication had to remain stable during the 14 weeks of the study.

Furthermore: schizophrenic disorder, a piece if metal in the brain, pacemaker and left-handed patients.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2004-05; Study Completion 2006-12

PRIMARY OUTCOMES:
To determine the depression (and so the effect of the treatment)we use the 10-item Montgomery Asberg Depression Rating Scale (MADRS)and we measure before tms (T=0), at week 1 (T=1), at week 2 (T=2), at week 4 (T=3), at week 8 (T=4), at week 14 (T=5)
Besides the MADRS we use the BDI (Beck depression Inventory, the Hamillton deppression and anxiety scale)

SECONDARY OUTCOMES:
-Changes in anxiety
-.Autonomic changes
-.changes in the emotioneal attention, in the emotional memory en in de emotional recognition.
-.Biochemical changes
-.Changes in the EEG
>> measured before tms and after (at T=0 and T=2)

CONTACTS AND LOCATIONS:
Overall Officials: G.F Koerselman, prof. dr., Study Director — st Lucas Andreas Ziekenhuis
Locations (1):
- st. Lucas Andreas Ziekenhuis/ Hospital, Amsterdam, Netherlands